CLINICAL TRIAL: NCT06193564
Title: Investigation of the Effects of Transcranial Direct Current Stimulation Combined With Stabilization Exercises on Functional Status, Cognitive Functions, and Sleep Quality in Individuals With Chronic Neck Pain: A Randomized Controlled Study
Brief Title: The Effects of tDAS Combined With Stabilization Exercises in Individuals With Chronic Neck Pain
Acronym: tDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, TDERE, Physiotherapist, Master Student (PT, MSc), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDERE; 1919B012105580 (Other Grant/Funding Number: THE SCIENTIFIC AND TECHNOLOGICAL RESEARCH COUNCIL OF TÜRKİYE)
Record Dates: First submitted 2023-12-10; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
Keywords: Transcranial direct current stimulation; neck pain; endurance; functional status; cognitive function
MeSH Terms: conditions — Neck Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined CSE with tDCS (Experimental): Combined cervical stabilzation exercises with tDCS
  Interventions: Other: Transcranial Direct Current Stimulation; Other: Cervical Stabilization Exercises
- control group (Experimental): Only cervical stabilzation exercises
  Interventions: Other: Cervical Stabilization Exercises
- placebo tDCS and CSE (Placebo Comparator): Placebo tDCS and cervical stabilzation exercises
  Interventions: Other: Cervical Stabilization Exercises; Other: Sham-Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) tDCS was administered using electrodes made of metal or conductive rubber, an electrode sponge, and an electrolyte-based contact medium applied to the sponge (6 ml of water for a 35 cm2 sponge). 'Chatanooga Ionto Iontophoresis Dual Channel System (USA)' was used in the study as a constant current stimulator for tDCS. The constant current stimulator was used to deliver the direct current in a constant manner by monitoring the resistance in the continuous system. Two electrodes were placed at 5 cm × 7 cm; 35 cm2; an anode was placed in the primary motor cortex (M1), while a cathode was placed in the contralateral supraorbital space (FP1 on the left and FP2 on the right, according to the EEG 10/20 system) A constant current of 2 mA was applied to the experimental group for 20 minutes.
  Arms: Combined CSE with tDCS
Other: Cervical Stabilization Exercises — Before initiating the stabilization exercises, individuals included in the study were instructed on correct postural alignment. Cervical chin tuck movement was taught during the exercise along with postural alignment and craniocervical flexion movement was requested. After teaching craniocervical flexion exercises in all positions (supine, lying on the side, prone, crawling, sitting, and standing), participants were instructed to perform the movement slowly.
  The purpose of this phase was to establish the relationship between vision and motor learning using the Pressure Biofeedback Stabilizer device. The device was positioned on the neck area and inflated to 20 mmHg. The pressure level gradually increased in 2-mmHg increments from 20 to 30 mmHg. For each pressure value (22, 24, 26, 28, 30 mmHg), participants were asked to maintain craniocervical flexion for 10 seconds, and this exercise was repeated ten times.
Other: Sham-Transcranial Direct Current Stimulation (tDCS) — tDCS was administered using electrodes made of metal or conductive rubber, an electrode sponge, and an electrolyte-based contact medium applied to the sponge (6 ml of water for a 35 cm2 sponge). 'Chatanooga Ionto Iontophoresis Dual Channel System (USA)' was used in the study as a constant current stimulator for tDCS. The constant current stimulator was used to deliver the direct current in a constant manner by monitoring the resistance in the continuous system. Two electrodes were placed at 5 cm × 7 cm; 35 cm2; an anode was placed in the primary motor cortex (M1), while a cathode was placed in the contralateral supraorbital space (FP1 on the left and FP2 on the right, according to the EEG 10/20 system) (Figure 2). As shown in the figure, a constant current of 2 mA was applied to the experimental group for 20 minutes. For the sham group, electrodes were placed in the same areas and a current of 0 mA was applied.
  Arms: placebo tDCS and CSE

SUMMARY:
The aim of study was to investigate the effect of cervical stabilization exercises (CSE) combined with tDCS on functional status, cognitive functions and sleep quality in individuals with chronic neck pain. A total of 29 individuals with chronic neck pain (33.06±14.81 age) were included in the study. Combined CSE with tDCS (2 mA/20 min) was applied to the experimental group (n=10); only CSE was applied to the control group (n=10); placebo tDCS (0 mA/20 min) and CSE were applied to the sham group (n=9). Before and after the 8-week intervention comprising a total of 16 sessions, the following assessments were carried out: Visual Analog Scale (VAS), Neck Bournemouth Questionnaire (NBQ), Cervical Muscle Endurance Tests, The Profile Fitness Mapping Neck Questionnaire (ProFitMap-neck), Montreal Cognitive Assessment (MoCA), Trail Making Test (TMT) and Pittsburgh Sleep Quality Index (PSQI).

DETAILED DESCRIPTION:
This study was conducted at Erciyes University Faculty of Sports Sciences with individuals suffering from chronic neck pain. The study included a total of 29 individuals with chronic neck pain, grouped into experimental, control, and sham groups. The flowchart in Figure 1 illustrates the distribution of individuals within each group.

The present study was conducted with individuals between 18 and 65 years of age who had suffered from neck pain for at least 3 months, with a rest pain score of 3-7 on the "Visual Analog Scale", without neurological deficits and without pathological findings (fractures, dislocations, tumors, infections) in radiological tests. In addition, neurological or psychiatric disorders, including acute/chronic depression, history of head trauma resulting in loss of consciousness, epilepsy, history of neurosurgical intervention, intracranial hypertension, implanted devices, history of migraine, history of chronic/severe headache, skin conditions (psoriasis, etc.), uncontrollable diseases (endocrinologic, cardiovascular, pulmonary, hematologic, hepatic, renal), presence of systemic inflammatory disease or malignancy, were excluded from the study.

Potential Confounders Gender, age, body mass index, smoking history, presence of back pain in the previous six months, chronic illness, and resting neck pain severity were considered potential confounders.

Study Design Cervical stabilization exercises (CSE) (20 min) with tDCS (2 mA) were administered to the experimental group of the study (n=10) for 20 min. Only CSE (20 min) was applied to the control group (n=10). To the Sham group (n=9); CSE (20 min) was administered with 20 min tDCS (0 mA). All cervical stabilization exercises were performed with a stabilizer biofeedback device (Stabilizer Pressure Biofeedback, Chattanooga Group Inc., USA) under the supervision of a physiotherapist. All groups were trained for a total of 16 sessions over 8 weeks (2 days/week).

Intervention Transcranial Direct Current Stimulation (tDCS) tDCS was administered using electrodes made of metal or conductive rubber, an electrode sponge, and an electrolyte-based contact medium applied to the sponge (6 ml of water for a 35 cm2 sponge). 'Chatanooga Ionto Iontophoresis Dual Channel System (USA)' was used in the study as a constant current stimulator for tDCS. The constant current stimulator was used to deliver the direct current in a constant manner by monitoring the resistance in the continuous system. Two electrodes were placed at 5 cm × 7 cm; 35 cm2; an anode was placed in the primary motor cortex (M1), while a cathode was placed in the contralateral supraorbital space (FP1 on the left and FP2 on the right, according to the EEG 10/20 system). As shown in the figure, a constant current of 2 mA was applied to the experimental group for 20 minutes. For the sham group, electrodes were placed in the same areas and a current of 0 mA was applied.

Cervical Stabilization Exercises Before initiating the stabilization exercises, individuals included in the study were instructed on correct postural alignment. Cervical chin tuck movement was taught during the exercise along with postural alignment and craniocervical flexion movement was requested. After teaching craniocervical flexion exercises in all positions (supine, lying on the side, prone, crawling, sitting, and standing), participants were instructed to perform the movement slowly.

The purpose of this phase was to establish the relationship between vision and motor learning using the Pressure Biofeedback Stabilizer device. The device was positioned on the neck area and inflated to 20 mmHg. The pressure level gradually increased in 2-mmHg increments from 20 to 30 mmHg. For each pressure value (22, 24, 26, 28, 30 mmHg), participants were asked to maintain craniocervical flexion for 10 seconds, and this exercise was repeated ten times.

Outcomes Measures After recording the demographics and information of all participants, we conducted the assessments below. All pre-treatment assessments were re-administered for the second time at the end of the 8-week training.

Assessment of Pain Severity In order to evaluate the pain intensity of individuals with chronic neck pain, 10-cm Visual Analogue Scale (VAS) developed by Price et al and the Neck Bournemouth Questionnaire (NBQ) developed by Bolton et al, were utilized. The 10-cm VAS is used to mark pain on a horizontal line where the first notch is 0, indicating no pain, and the last notch is 10, indicating the most severe pain. Participants marked their neck pain levels on the line, and the measurements were recorded in centimeters using a ruler. The NBQ was used to inquire about participants' neck pain severity as well as symptoms such as the impact of neck pain on their daily activities and social life, levels of anxiety and depression, kinesiophobia, and methods of coping with pain in the previous week. The Turkish version of the NBQ, validated for reliability by Telci et al, consists of 7 questions, each scored on a scale of 0 to 10. A possible total score of 70 indicates more severe neck pain.

Assessment of Functional Status Assessment of Muscular Endurance To evaluate the cervical deep flexor muscular endurance test, participants took a hook-lying posture on a therapy table, maintaining a neutral neck position with the head and neck straightly aligned. With the assistance of a stabilizing device, a pressure sensor was situated under the neck with a stabilizer (Stabilizer Biofeedback). Participants were instructed to simulate a "yes" motion by gently nodding their heads, while avoiding movements that could activate the sternocleidomastoid muscle. The test involved a pressure range of 20-30 mmHg and required ten-second sustained pressure at each 2-mmHg increment without any breaks. The activation score was determined by measuring the pressure level at which the patient was able to perform and sustain 10 repetitions for a duration of 10 seconds, providing a measure of the strength of the deep cervical flexor muscles. The endurance performance index was determined by analyzing the number of successful repetitions completed by the patient while maintaining a constant pressure level for a duration of 10 seconds. The maximum activation score was 10 mmHg, and the maximum performance index was 100. To assess the endurance of neck extensor muscles, participants were given a 2-kg weight attached to the C6 level using a 10-centimeter velcro while lying prone. Their hands were placed on both sides, and the maximum duration they sustained their head in that position was recorded in seconds. The study assessed the endurance of cervical flexor muscles in participants with chronic neck pain. Participants positioned themselves in a supine hooked position, with their hands on the abdomen and chin retracted. The maximum time a participant could raise and sustain their head at a height of approximately 2.5 cm was noted in seconds.

Assessment of Functional Limitations and Symptoms The Profile Fitness Mapping neck questionnaire (ProFitMap-neck) was used to assess the functional limitations and symptoms associated with neck pain. The survey was graded on a scale of 0-100%, showing the highest score possible. This was the best result attainable through the assessment of the questionnaire. In addition to assessing neck pain, ProFitMap-neck considers stiffness, tension, and weakness that might occur in the neck and hands. This survey consists of two sub-indices. The first consists of 26 items that comprehensively assess the frequency and severity of symptoms, while the second comprises 18 items that assess functional limitations. Symptom frequency is rated on a scale of 1 to 6 points, where 1 indicates "not at all/rarely" and 6 corresponds to "often/always," as described in the Symptom Frequency Index. Symptom severity was rated on a scale of 7 to 12, with 7 being "not at all" and 12 being "almost unbearable/unbearable/very severe/extreme," based on the Symptom Severity Index. Individuals rated their experiences on a scale of 1 to 6, where 1 was "very good/no problem/no disturbance" and 6 was "very bad/very difficult/disturbing/impossible," according to the Functional Limitation Index. The reliability of the questionnaire in the Turkish context was validated by Çetin et al.

Assessment of Cognitive Status Individuals' cognitive status was assessed using the Montreal Cognitive Assessment (MoCA). The MoCA is a concise measurement tool developed by Ziad Nasreddine et al and used to detect mild cognitive impairment. The MoCA score ranges from 0 to 30, and 26 points and above is considered as a normal cognitive function. The Turkish version of the MoCA, in which cultural and linguistic adaptations were made, was used for the cognitive function of participants. The scale evaluates seven cognitive domains including attention, concentration, executive functions, memory, language, visual construction skills, abstract thinking, calculation, and orientation. The domains assess various cognitive abilities through tasks. Participants who scored 21 and above out of 30 points were in the normal group. The test took an average of 10 minutes to complete.

The Trail Making Test is a cognitive assessment tool that evaluates various cognitive functions such as visual-motor coordination, conceptual scanning, motor speed, planning, numerical knowledge, abstract thinking, and response tendency based on physical attributes of stimuli, set shifting, concentration, and tolerance to interference. It consists of two parts, referred to as Part A and Part B. Part A uses numbers as stimuli, and the participant's task is to connect the numbered circles in the correct order (1-2-3-4-5...) without interruption. Part B consists of circles that contain both letters and numbers. To complete this task, participants are asked to connect the circles by drawing straight lines, alternating between numbers and letters in a sequential order (1-A-2-B-3-C-4-D...). A normative study conducted by Türkeş et al verified that the Trail Making Test (TMT) is reliable for the Turkish population. In the study, the original versions of Part A and Part B of the Trail Making Test will be utilized.

Assessment of Sleep Quality The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality in individuals with chronic neck pain. The PSQI utilizes a standardized questionnaire to distinguish between good and poor sleepers. This comprises 19 self-rated questions and 5 questions answered by a bedmate/roommate. These 5 questions do not contribute to the scoring from a clinical perspective. The items of the PSQI use various response categories, including recording usual bedtime, usual wake time, number of hours actually slept, and number of minutes to fall asleep, as well as forced-choice Likert-type responses (0-3). The total scores of the components generate a single global score, ranging from 0 to 21. Higher scores indicate poorer sleep quality. In a study conducted in Turkey by Ağargün et al, it was established that a global PSQI score greater than 5 indicates poor sleep quality. Buysse et al also reported good internal consistency (α = 0.83) and test-retest reliability (r = 0.85), with a total score of 8.0 or higher indicating subpar sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 65 years of age who had suffered from neck pain for at least 3 months
* The rest pain score of 3-7 on the "Visual Analog Scale" (Javdaneh et al, 2021)

Exclusion Criteria:

* Neurological or psychiatric disorders,
* including acute/chronic depression, history of head trauma resulting in loss of consciousness
* epilepsy
* history of neurosurgical intervention
* intracranial hypertension
* implanted devices
* history of migraine
* history of chronic/severe headache
* skin conditions (psoriasis, etc.), uncontrollable diseases (endocrinologic, cardiovascular, pulmonary, hematologic, hepatic, renal)
* presence of systemic inflammatory disease or malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain Severity | January 2023 to November 2023 (10 months)
  In order to evaluate the pain intensity of individuals with chronic neck pain, 10-cm Visual Analogue Scale (VAS) developed by Price et al. The 10-cm VAS is used to mark pain on a horizontal line where the first notch is 0, indicating no pain, and the last notch is 10, indicating the most severe pain. Participants marked their neck pain levels on the line, and the measurements were recorded in centimeters using a ruler.
Assessment of Pain Severity | January 2023 to November 2023 (10 months)
  The NBQ was used to inquire about participants' neck pain severity as well as symptoms such as the impact of neck pain on their daily activities and social life, levels of anxiety and depression, kinesiophobia, and methods of coping with pain in the previous week. The Turkish version of the NBQ, validated for reliability by Telci et al, consists of 7 questions, each scored on a scale of 0 to 10. A possible total score of 70 indicates more severe.
Assessment of Muscular Endurance | January 2023 to November 2023 (10 months)
  To evaluate the cervical deep flexor muscular endurance test, participants took a hook-lying posture on a therapy table, maintaining a neutral neck position with the head and neck straightly aligned. With the assistance of a stabilizing device, a pressure sensor was situated under the neck with a stabilizer (Stabilizer Biofeedback). Participants were instructed to simulate a "yes" motion by gently nodding their heads, while avoiding movements that could activate the sternocleidomastoid muscle. The test involved a pressure range of 20-30 mmHg and required ten-second sustained pressure at each 2-mmHg increment without any breaks. The activation score was determined by measuring the pressure level at which the patient was able to perform and sustain 10 repetitions for a duration of 10 seconds, providing a measure of the strength of the deep cervical flexor muscles.
Assessment of Functional Limitations and Symptoms | January 2023 to November 2023 (10 months)
  The Profile Fitness Mapping neck questionnaire (ProFitMap-neck) was used to assess the functional limitations and symptoms associated with neck pain. The survey was graded on a scale of 0-100%, showing the highest score possible. This was the best result attainable through the assessment of the questionnaire. In addition to assessing neck pain, ProFitMap-neck considers stiffness, tension, and weakness that might occur in the neck and hands. This survey consists of two sub-indices. The first consists of 26 items that comprehensively assess the frequency and severity of symptoms, while the second comprises 18 items that assess functional limitations. Symptom frequency is rated on a scale of 1 to 6 points, where 1 indicates "not at all/rarely" and 6 corresponds to "often/always," as described in the Symptom Frequency Index. Symptom severity was rated on a scale of 7 to 12, with 7 being "not at all" and 12 being "almost unbearable/unbearable/very.
Assessment of Cognitive Status | January 2023 to November 2023 (10 months)
  Individuals' cognitive status was assessed using the Montreal Cognitive Assessment (MoCA). The MoCA is a concise measurement tool developed by Ziad Nasreddine et al and used to detect mild cognitive impairment. MoCA application takes approximately 10 minutes. The highest total score that can be obtained from the test is 30. Accordingly, a score of 21 points or above is considered normal.
Assessment of Cognitive Status | January 2023 to November 2023 (10 months)
  The Trail Making Test is a cognitive assessment tool that evaluates various cognitive functions such as visual-motor coordination, conceptual scanning, motor speed, planning, numerical knowledge, abstract thinking, and response tendency based on physical attributes of stimuli, set shifting, concentration, and tolerance to interference. Scoring is based on time taken to complete the test (e.g. 35 seconds yielding a score of 35) with lower scores being better. Different norms are available that allow comparison with age-matched groups.
Assessment of Sleep Quality | January 2023 to November 2023 (10 months)
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality in individuals with chronic neck pain. The PSQI utilizes a standardized questionnaire to distinguish between good and poor sleepers. This comprises 19 self-rated questions and 5 questions answered by a bedmate/roommate. These 5 questions do not contribute to the scoring from a clinical perspective. The items of the PSQI use various response categories, including recording usual bedtime, usual wake time, number of hours actually slept, and number of minutes to fall asleep, as well as forced-choice Likert-type responses (0-3). The total scores of the components generate a single global score, ranging from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba DERE, Principal Investigator — Yozgat Bozok University
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University, Talas, Kayseri
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iqbal ZA, Alghadir AH, Anwer S. Efficacy of Deep Cervical Flexor Muscle Training on Neck Pain, Functional Disability, and Muscle Endurance in School Teachers: A Clinical Trial. Biomed Res Int. 2021 Jan 13;2021:7190808. doi: 10.1155/2021/7190808. eCollection 2021. PMID 33521131
- [Result] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Result] Juan W, Rui L, Wei-Wen Z. Chronic neck pain and depression: the mediating role of sleep quality and exercise. Psychol Health Med. 2020 Sep;25(8):1029-1035. doi: 10.1080/13548506.2020.1724308. Epub 2020 Feb 4. PMID 32013565